CLINICAL TRIAL: NCT05155735
Title: Functional Outcomes of Single Digit Replantation Versus Revision Amputation, a Prospective Study
Brief Title: Functional Outcomes of Single Digit Replantation Versus Revision Amputation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-10233
Record Dates: First submitted 2021-11-01; First posted 2021-12-14 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Amputation; Traumatic, Hand
Keywords: Replantation; Single digit; function; DASH
MeSH Terms: interventions — Replantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Replantation: This group will include subjects who suffered a single digit non-thumb amputation, and whose finger was replanted.
  Interventions: Procedure: Replantation
- Revision Amputation: This group will include subjects who suffered a single digit non-thumb amputation, and whose finger was not replanted.
  Interventions: Procedure: Primary wound closure

INTERVENTIONS:
Procedure: Replantation — Surgical reattachment of a severed body part
  Groups: Replantation
Procedure: Primary wound closure — Primary wound closure with removal of exposed bone
  Groups: Revision Amputation

SUMMARY:
The purpose of this study is to compare functional outcomes in single digit replantation subjects compared with revision amputation. Functional outcomes will be assessed by DASH (disabilities of the arm, shoulder and hand) score and with Purdue Pegboard Test by the subject's respective hand therapist at their last visit. Results will contribute to generating a preoperative decision algorithm for single digit amputation injuries.

DETAILED DESCRIPTION:
Research design: Prospective observational cohort study

Study population, enrollment, and duration of participation:

Collaborating institutions Revision amputation cohort: CHUM, Santa Cabrini Hospital and Maisonneuve Rosemont Hospital Replantation cohort: CEVARMU/CHUM

Inclusion Criteria: All replantation and revision amputation of single digits who are treated at the collaborating hospital centres Exclusion Criteria: Thumb amputation, Multiple digit amputation, Failure to follow-up with an occupational therapist

Enrollment:

Database encompassing regional plastic surgery interventions will be reviewed to target patients who underwent single digit replantation and revision amputation in the last year, up until the first patient that is not scheduled to come back for evaluation with his hand therapist (as not to introduce a selection bias). Going forward we will run prospectively until we have sufficient data to yield significant results, as the rarity of single digit replantation will be the limiting factor. On call plastic surgery residents at our institution will also be advised to contact the research personnel when they encounter possible candidates at the participating hospitals. The research personnel will in no instance intervene nor influence the decision-making process leading to either revision amputation or replantation of the single digit. Post-operatively, the research personnel will review the patient files to select participants meeting the selection criteria.

Participants will be classified to the following groups according to the intervention performed:

* Replantation group
* Revision amputation group
* Crossover group (initially replanted, then underwent revision amputation) Subgroups
* Injured digit (index, middle, ring, little)
* Injury level: Tamai classification

  * Zone 1 (distal to FDP insertion)
  * Zone 2 (distal to interphalangeal joint until FDP insertion)
  * Zone 3 (middle phalanx distal to FDS insertion)
  * Zone 4 (proximal phalanx until middle phalanx FDS insertion) o Zone 5 (metacarpophalangeal joint and proximal)
* Mechanism of injury o Guillotine

  * Minor crush
  * Major crush o Avulsion

The following data will be retrieved from the patients filles:

Demographic variables/Patient characteristics

* Age
* Gender
* Smoking status: cigarette and cannabis
* Patient comorbidity:

  * Diabetes mellitus
  * Hypertension
* Hand dominance
* Patient preference: cultural beliefs Variables possibly influencing outcome
* Ischemia time
* Workers' compensation
* Revision surgery
* Acute post-op complications o Infection

  * Bleeding
  * Vascular thrombosis o Other
* Chronic complications o Tendon rupture

  * Tendon adhesions
  * Bony malunion
  * Bony non-union
  * Painful neuroma formation o CRPS
  * Other

Evaluation phase and follow-up Each patient's respective hand therapist will then be contacted to be introduced to the research protocol. Instructions regarding patient consent and evaluation tools will be explained. Hand therapists who have the necessary materials and tools to administer the tests and who are willing to participate in the study will receive a copy of the research protocol, detailed instructions regarding their participation and the consent form.

End-of-hand therapy is defined as the last or second-to-last follow-up appointment with the collaborating hand therapist. At this moment, the hand therapist will introduce the patient to the research protocol and will obtain their informed written consent. The DASH score (appendix 1) will then be administered by the occupational therapist in a standardized manner to all participants. Lastly, a quantitative hand function test will be conducted using the Purdue Pegboard according to the standardized procedure described in the user manual by Lafayette Instrument Company, Inc. Both the injured and the non-injured hand will be tested.

A secured online excel sheet will be shared amongst all the collaborating occupational therapists to record the test results.

Statistical Methods:

In order to detect a significant difference in average functional outcome between the two study groups, we will conduct a two-sided t-test using the SPSS software (IBM SPSS, V26, NY). By choosing our cut-off to be 0.05 and a beta of 0.1, we gained 90% power (1 - beta), accordingly we will deem a p-value of ≤ 0.05 as statistically significant. Continuous data will be expressed as mean and standard deviation or median and range, and assessed with t test. Categorical (nominal) data will be summarized as the frequency (%) and we will utilize Pearson Chi-Square and Fisher's exact tests for analysis. We then will analyze the outcomes by logistic regression model comprising two study groups, sex, patient's comorbidities and habit of smoking, and the mechanism of injury. Multiple linear regression analysis will be performed to measure and control confounding variables.

Results obtained from the study will then be used to generate a preoperative decision algorithm for single digit replantation vs. revision amputation. This could help guide clinicians from peripheral centres with questions about medico-legal issues.

Safety Management:

Since the study procedures are not greater than minimal risk, serious adverse events (SAE) are not expected. If any unanticipated problems related to the research involving risks to subjects or others happen during the course of this study (including SAEs) these will be reported to the IRB in accordance with the procedure described in the Mode opératoire normalisé-10: Gestion des évènements indésirables. Adverse events (AEs) that are not serious but that are notable and could involve risks to subjects will be summarized in narrative or other format and submitted to the CÉR at the time of continuing review.

ELIGIBILITY:
Inclusion Criteria:

* Replantation of single digits treated at collaborating hospital centres
* Revision amputation of single digits treated at collaborating hospital centres

Exclusion Criteria:

* Thumb amputation
* Multiple digit amputation
* Failure to follow-up with hand therapist

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects who have suffered a single digit amputation who are treated at the collaborating hospital centres
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Functional outcome by DASH score | Immediately following patient discharge from hand therapy
  Measured by DASH score (higher scores indicate a greater level of disability, score range from 0 to 100)
Functional outcome by Purdue Pegboard Test | Immediately following patient discharge from hand therapy
  Measured by Purdue Pegboard Test (higher scores indicate a greater level of dexterity and functionality and are typically compared with normative data stratified on the basis of age, score range depends on how the test is administered)
Functional outcome by Michigan Hand Questionnaire | Immediately following patient discharge from hand therapy
  Measured by Michigan Hand Questionnaire (higher scores indicate a greater level of functionality, score range from 0 to 100)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Mastropasqua, MD, Principal Investigator — Université de Montréal
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal East, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stone N, Shah A, Chin B, McKinnon V, McRae M. Comparing digital replantation versus revision amputation patient reported outcomes for traumatic digital amputations of the hand: A systematic review and meta-analysis. Microsurgery. 2021 Jul;41(5):488-497. doi: 10.1002/micr.30738. Epub 2021 Apr 3. PMID 33811398
- [Background] Kaplan FT, Raskin KB. Indications and surgical techniques for digit replantation. Bull Hosp Jt Dis. 2001-2002;60(3-4):179-88. PMID 12102407
- [Background] Tejedor Navarro A, Vendrell Jorda M, Puente Alonso C. Digital replantation/revascularization: predictive factors to microsurgery success-a single-center study. Eur J Trauma Emerg Surg. 2021 Feb;47(1):225-232. doi: 10.1007/s00068-019-01226-x. Epub 2019 Sep 24. PMID 31552437
- [Background] Zhu H, Bao B, Zheng X. A Comparison of Functional Outcomes and Therapeutic Costs: Single-Digit Replantation versus Revision Amputation. Plast Reconstr Surg. 2018 Feb;141(2):244e-249e. doi: 10.1097/PRS.0000000000004024. PMID 29036026
- [Background] Shaterian A, Sayadi LR, Tiourin E, Gardner DJ, Evans GRD, Leis A. Predictors of Hand Function Following Digit Replantation: Quantitative Review and Meta-Analysis. Hand (N Y). 2021 Jan;16(1):11-17. doi: 10.1177/1558944719834658. Epub 2019 Apr 2. PMID 30938181